CLINICAL TRIAL: NCT05910619
Title: Transcranial Pulse Stimulation of the Brain in Older Adults With and Without Mild Dementia
Brief Title: Transcranial Pulse Stimulation of the Brain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202300156
Record Dates: First submitted 2023-06-06; First posted 2023-06-20 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Mild Dementia; Aging Well
Keywords: Mild Dementia; Typical Aging; Transcranial Pulse Stimulation

STUDY DESIGN:
Intervention Model Description: 2x2 sham-controlled design in which 10 typically-aging older adults and 10 patients with mild AD will be randomized to receive either sham TPS or active TPS
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All parties involved will be blinded to the participant condition with the exception of 1) the interventionist applying the pulsed stimulation to the participant brain, as they will be required to ensure the TPS device is set to sham/active before application of the stimulation, and 2) the biostatistician who will randomize participants with sex-stratification
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active brain stimulation (Active Comparator): These participants will receive focused TPS (pulsed stimulation) of the specified default mode network regions as specified in the detailed study description.
  Interventions: Device: Neurolith Transcranial Pulse Stimulation Active
- Sham brain stimulation (Sham Comparator): These participants will also receive focused TPS (pulsed stimulation) of the specified default mode network regions as specified in the detailed study description, though the device will be set to "Sham" in a blinded fashion by the biostatistician by placing an air pouch in the device hand piece.
  Interventions: Device: Neurolith Transcranial Pulse Stimulation Sham

INTERVENTIONS:
Device: Neurolith Transcranial Pulse Stimulation Active — 5hz (200-300 milliseconds) stimulation pulses transcranial pulse stimulation (TPS) will be applied to each of the following five regions twice per session in sequential order with the specified stimulation parameters: left dorsolateral prefrontal cortex and inferior frontal cortex extending to Broca's area (2x800 pulses), right dorsolateral prefrontal cortex and inferior frontal cortex extending to Broca's area (2x800 pulses; ROI volume ~136/164 cms), the left lateral parietal cortex extending to Wernicke's area (2x400 pulses; ROI volume ~122/147 cms), the right lateral parietal cortex extending to Wernicke's area (2x400 pulses; ROI volume ~122/147 cms), and the extended precuneus cortex (2x600 pulses; ROI volume 66/92 cms). With a repetition time of 5hz (0.00333 seconds) per pulse at a total of 6,000 pulses per participant, the duration of stimulation is about 20 minutes, not including transition time between ROI localization.
  Arms: Active brain stimulation
Device: Neurolith Transcranial Pulse Stimulation Sham — The intervention procedure described in the Active condition above will also be repeated in participants randomized to the Sham procedure, with the exception of the insertion of a lens over the device by the interventionist to prevent stimulation from reaching the brain.
  Arms: Sham brain stimulation

SUMMARY:
This study will investigate transcranial pulse stimulation (TPS) as a method of enhancing cognitive and neural function. The study team will apply this low intensity, magnetically pulse technology to key brain regions in a randomized, sham-controlled trial (RCT). The study will determine the magnitude of changes in cognitive function and brain function and structure between a pre- and post-stimulation among 10 typically-aging older adults and 10 patients with mild dementia.

DETAILED DESCRIPTION:
The current study will investigate the use of the NEUROLITH TPS (transcranial pulse stimulation) generator device (Storz Medical AG, Tägerwilen, Switzerland) for enhancing cognitive and neural function in older adults with and without mild Alzheimer's disease (AD). This will be achieved by applying a novel, low intensity, magnetically pulsed technology to key brain regions and networks in a randomized, sham-controlled trial (RCT). The pilot RCT will be conducted to determine the magnitude of changes in cognitive function and brain function and structure between a pre- and post-stimulation using a 2x2 sham-controlled design in which 10 typically-aging older adults and 10 patients with mild AD will be randomized to receive either sham TPS or active TPS. All participants will undergo pre-intervention multi-modal MRI, blood draw, and neurocognitive evaluation followed by thrice-weekly TPS (sham or active) for two weeks total, followed by a post-intervention MRI, blood draw, and neurocognitive evaluation. The total duration of the study is expected to be around four weeks, where each participant will undergo a screening/eligibility visit, baseline visit with MRI and neurocognitive testing, 6 intervention visits, a post-intervention MRI and neurocognitive testing visit after the final stimulation session for a total of about 9 in-person visits. The final week of the study is a no-contact period in which the participant will be called approximately seven days after their final stimulation session to ensure no adverse events have occurred. The team will also contact participants quarterly for one year after the final session to complete a five minute phone survey.

The central hypothesis of this proposal is that TPS will increase cortical thickness, cerebral blood flow, neurite orientation and dispersion, and functional connectivity in targeted regions and their associated networks. Further, we hypothesize that these changes will translate to improvements in neurocognitive function more than that seen in the sham intervention, which is likely to occur due to practice effects alone.

The objectives of this study are to:

Aim 1. Determine whether application of TPS is associated with neurocognitive improvement H1.1. For both typically-aging older adults and patients with mild AD, active TPS will result in greater neurocognitive gains than sham TPS on a primary outcome measure of global cognition obtained from the ADAS-Cog-plus battery.

H1.2. Neurocognitive gains on the recall memory measures in active TPS will be greater for patients with mild AD compared to typically-aging older adults.

Aim 2. Determine whether TPS leads to improvements in functional (rsfMRI, ASL) and structural brain changes (NODDI).

H2.1. Active TPS targeting the AD-relevant regions and networks will potentiate increased connectivity in attention and working memory related (dorsolateral prefrontal cortex) brain systems, reflecting increased neural efficiency, while sham TPS will not.

H2.2. Active TPS will result in increased cerebral blood flow in targeted regions compared to sham TPS as measured by change in arterial spin labeling (ASL) metrics.

H2.3. White matter integrity will remain stable in the active TPS condition, with stable neurite density and neurite orientation dispersion occurring in targeted regions.

Aim 3. Evaluate which baseline neuroimaging characteristics best predict treatment response H3.1. In both typically aging older adults and mild AD, baseline within-network connectivity of the default mode network will be positively associated with change in a secondary outcome measure of executive function (NIH Examiner) for those randomized to active TPS, but not in sham TPS.

H3.2. In mild AD, average baseline neurite density within the white matter of the targeted regions will be positively associated with change in ADAS-Cog-plus total score after active TPS.

Exploratory Aim. Determine whether the intervention results in a clinically meaningful change in blood (plasma) based AD-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age: 65 to 84 years
* English speaking
* Physically mobile with no history of balance difficulties or major falls
* For the typically-aging older adult group, phone screening performance on the TICS must be greater than or equal to 33 points, and cognitive performance of 26 points or greater on the MoCA and a Sum of Boxes score of 0 on the Clinical Dementia Rating scale administered to the participant's informant at the initial visit
* For the Mild dementia group, phone screening performance on the TICS must be between 21 and 32 points, and subsequent cognitive performance of on the MoCA must be <23 with a CDR Sum of Boxes score between 4.5 and 9.0 as administered to the participants known informant at the initial visit.

Exclusion Criteria:

* Neurological disorders unrelated to dementia / AD (e.g., Parkinson's disease, stroke, seizures, traumatic brain injury)
* Evidence of greater-than-mild dementia/AD (based on informant CDR Sum of Boxes score greater than 9.0 or MoCA <10)
* Past opportunistic brain infection
* Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis or severe major depression and/or suicidality) or any history of agitation and/or delirium
* Unstable (e.g., cancer other than basal cell skin) and chronic (e.g., diabetes mellitus) medical conditions
* MRI contraindications (e.g., pregnancy, claustrophobia, metal implants that are contraindicated for MRI and TPS)
* Physical impairment precluding motor response or lying still for one hour and inability to walk two blocks without stopping or without balance difficulties
* Drug exclusions include those medications that are known to have cognitively sedating or altering effects as well medications with a strong anticholinergic burden or CNS effects. Participants should be stable on any recently altered medications/dosages for at least four weeks prior to beginning the study. Medications will be reviewed during the interview for the purpose of identification of contraindicated pharmacological agents with common cognitive side-effects
* Other history of medical conditions that may increase risk of cerebrovascular events, including prior heart attack, cardiac arrhythmia such as atrial fibrillation
* Hearing or vision deficits that will not allow for reliable standardized cognitive assessment; i.e. colorblindness, inability to hear through headphones (with or without hearing aids), macular degeneration or other significant diseases that cause severe loss of vision. If vision is corrected with lenses to appropriate levels, then participant will be eligible
* Left-handedness and ambidextrousness, as these individuals have a higher percentage rate of atypical functional lateralization for brain functions, which would significantly interfere with interpretability of brain data
* Hemophilia or other blood clotting disorders or thrombosis
* Corticosteroid treatment within the last six weeks before the first treatment

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
ADAS-Cog-Plus-EF&FA Battery Total Score | Four weeks
  The ADAS-Cog-Plus total score is touted as the gold standard measure for outcomes measurement following anti-dementia interventions18, allows for reliable longitudinal data collection, and provides coverage of cognitive domains including orientation, memory, language, and praxis.

SECONDARY OUTCOMES:
NIH Examiner Total Score | Four weeks
  The Total Score from the NIH Examiner will provide coverage of frontal executive functions in a manner that could be completed in a short time frame to limit participant burden. The NIH Examiner was chosen as it 1) Can be completed in ~30 minutes; 2) Is computerized and well standardized with norms from a large national cohort of older adults; 3) Provides both accuracy and response time measures; 4) Emphasizes working memory and executive function domains of relevance to the study which are not fully assessed by the ADAS-cog-plus battery; and 5) Has been the subject of considerable focus and investment by NIA.

OTHER OUTCOMES:
Arterial Spin Labeling MRI Cerebral Bloodflow Change | Four weeks
  Net change in cerebral blood flow of the targeted Default Mode Network regions after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gullett, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No